CLINICAL TRIAL: NCT01323062
Title: A Phase 1b Study of Bavituximab Plus Carboplatin and Pemetrexed in Chemotherapy-Naive Stage IV Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Bavituximab Plus Carbo and Pemetrexed in Chemo-Naive Stage IV Non-Squamous Non-Small Cell Lung Cancer (NSCLC) Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1030
Record Dates: First submitted 2011-03-08; First posted 2011-03-25 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: chemotherapy naive; stage IV non squamous non small cell lung cancer; Phase 1b; Bavituximab; Chimeric 3G4; U of North Carolina at Chapel Hill
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — bavituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-arm trial (Other): Single-arm trial
  Interventions: Drug: Bavituximab

INTERVENTIONS:
Drug: Bavituximab — Administered 3 mg/kg weekly
  Other Names: chimeric 3G4

SUMMARY:
This is a non-randomized, open-label Phase 1b trial to establish the safety and recommended phase 2 dose (RP2D) of bavituximab in combination with pemetrexed and carboplatin in subjects with previously untreated stage IV non-squamous non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Subjects with measurable disease will be assessed for response after every 2 cycles of therapy using RECIST 1.1 criteria. In addition, progression free survival (PFS), overall survival (OS) and exploratory biomarkers, imaging, and thrombotic risk parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18
* Histologically or cytologically confirmed stage IV non-squamous NSCLC not previously treated with systemic chemotherapy
* Evaluable disease by clinical or radiographic parameters
* No history or concomitant malignancy
* Adequate organ and marrow function
* Female subjects with negative urine or serum pregnancy
* ECOG must be 0 or 1

Exclusion Criteria:

* Squamous cell, small cell, or mixed histology
* Known history of bleeding diathesis or coagulopathy
* Cavitary tumors or tumors invading or abutting large blood vessels
* Any history of thromboembolic events
* Ongoing therapy with oral or parenteral anticoagulants
* Major surgery within 4 weeks of Day 1 of treatment
* Uncontrolled intercurrent disease (diabetes, hypertension, thyroid disease)
* any history of significant vascular disease
* Congestive heart failure
* History of any condition requiring anti-platelet therapy
* Serious non healing wound
* Known chronic infection with human immunodeficiency virus (HIV) or viral hepatitis
* Unable or unwilling to discontinue use of prohibited medications
* D-dimers >2 x ULN as measured on 2 separate occasions at least 1 day apart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05-14 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Measure number of severe side effects seen during first cycle of therapy | Three weeks
  To determine the maximum tolerated dose based on occurrence of dose-limititing toxicity (DLT) within the first 3 weeks of treatment to determine appropriate and safe dose of bavituximab in combination with carboplatin and pemetrexed

SECONDARY OUTCOMES:
Progression free survival | At the time from the start of treatment until documented disease as defined bia RECIST 1.1 or death
  to determine the overall response rate and estimate progression free survival associated with bavituximab in combination with carboplatin and pemetrexed

CONTACTS AND LOCATIONS:
Overall Officials: Juneko Grilley Olson, MD, Principal Investigator — U of North Carolina at Chapel Hill
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- See also: web address for Lineberger Comprehensive Cancer Center, UNC — http://www.unclineberger.org
- See also: web address for the National Cancer Institute (NCI) — http://www.cancer.gov